CLINICAL TRIAL: NCT01462214
Title: Phase 1-2 Study of Everolimus and Low-dose Cyclophosphamide in Patients With Metastatic Renal Cell Cancer.
Brief Title: Study of Everolimus and Low-dose Cyclophosphamide in Patients With Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hans J. van der Vliet, MD, PhD (Other)
Collaborators: Dutch Cancer Society (Other); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Hans J. van der Vliet, MD, PhD, Medical Oncologist, Department of Medical Oncology, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/016
Record Dates: First submitted 2011-10-10; First posted 2011-10-31 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Everolimus — Patients will be treated with low-dose oral cyclophosphamide (8 different dose levels and schedules) in combination with fixed dose (10 mg) everolimus in patients with mRCC.

SUMMARY:
In the present phase 1-2 study the investigators aim to determine whether depletion of Tregs using metronomic cyclophosphamide can enhance the antitumor efficacy of everolimus in patients with mRCC not amenable to or progressive after a VEGF-receptor tyrosine kinase inhibitor containing treatment regimen. In the phase 1 part of the study the investigators will determine the optimal CD4+CD25+ regulatory T cell-depleting dose and schedule of metronomic oral cyclophosphamide when given in combination with a fixed dose (10 mg daily) of everolimus. In the phase 2 part of the study the investigators will subsequently evaluate whether the number of patients who are cancer progression free at 4 months can be increased from 50% to 70% by adding metronomic cyclophosphamide (in the dose and schedule determined in the phase 1 part) to everolimus. In addition to efficacy, the investigators will evaluate treatment toxicity to determine whether this combination strategy is feasible and safe.

DETAILED DESCRIPTION:
This is a phase I/II, national multi-center study of different doses and schedules of low-dose oral cyclophosphamide in combination with fixed dose everolimus in patients with mRCC not amenable to or progressive after a VEGF-receptor tyrosine kinase inhibitor containing treatment regimen. Phase I part: Patients will be enrolled in cohorts of 5 per dose level. The first 5 patients enrolled will be assigned to dose level 0 in order to assess immune and angiogenic effects caused by everolimus monotherapy. The second 5 patients enrolled will be assigned to dose level 1. If there are ≤1 dose-limiting toxicities (DLTs) experienced by the first 5 patients in a cohort during the first 28 days after the first study treatment, further patients will be entered in the next dose level. Entry of patients into the expansion cohort will not occur until at least 28 days after the last patient in the escalation phase received his/her first study treatment. At the final dose level recommended for the phase II study a minimum of 10 patients will be treated. Phase II part: In the phase 2 part of the study up to 56 patients will be treated at the dose level that has been selected based on its capacity to most selectively deplete circulating Treg levels in the phase 1 part of the study. Based on data of patients with mRCC treated with everolimus monotherapy after previous treatment with sunitinib ± sorafenib, the investigators aim to increase the number of patients who are alive and cancer progression free at 4 months from 50% to 70% by adding metronomic cyclophosphamide. In addition, the investigators consider this increase meaningful as long as the combination treatment does not cause combination treatment related toxicity ≥ grade 3 in ≥ 30% of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed clear-cell mRCC with progressive disease and not amenable to or progressive on or within 6 months of stopping treatment with a VEGF receptor tyrosine kinase inhibitor (sunitinib (or pazopanib) ± sorafenib).
* Prior therapy with cytokines (i.e. IL-2, interferon) and/or VEGF-ligand inhibitors (i.e. bevacizumab) is permitted.
* Patients with brain metastases are eligible if they have been stable for at least two months post-radiation therapy or surgery.
* Aged 18 years or older.
* No other current malignant disease, except for basal cell carcinoma of the skin.
* WHO performance status 0-2.
* Life expectancy of at least 12 weeks.
* Adequate hematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, Hb ≥ 6.0 mmol/L.
* Adequate hepatic function: serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5 x ULN (or ≤ 5 times ULN if liver metastases are present).
* Adequate renal function: calculated creatinine clearance ≥ 50 ml/min.
* Measurable or evaluable disease as defined by RECIST 1.1.
* Patients with reproductive potential must use effective contraception. Female patients must have a negative pregnancy test.
* Signed informed consent.
* Able to receive oral medication.

Exclusion Criteria:

* Patients currently receiving chemotherapy, immunotherapy, or radiotherapy or who have received these ≤ 4 weeks prior to visit 1. The wash-out period for sunitinib or sorafenib is at least 2 weeks from the first dose of the study medication.
* Known human immunodeficiency virus (HIV) or other major immunodeficiency.
* Immunosuppressive agents within 3 weeks of study entry, except for low dose corticosteroids when given for disorders such as rheumatoid arthritis, asthma, or adrenal insufficiency. Topical or inhaled corticosteroids are permitted.
* Patients with an active bleeding diathesis or on oral anti-vitamin K medication.
* Patients with untreated CNS metastases with clinical symptoms or who have received treatment for CNS metastases within 2 months of study entry. Patients with treated CNS metastases, who are neurologically stable and off of corticosteroids for more than 2 months prior to study entry are eligible to enter the study.
* Active infection or serious intercurrent illness, except asymptomatic bacteriuria.
* Presence of unstable angina, recent myocardial infarction (within the previous 6 months), or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia.
* Macroscopic hematuria
* Prior therapy with mTOR inhibitors. 10. Known hypersensitivity to everolimus or other rapamycins (sirolimus/temsirolimus) or to its excipients.
* Pregnant or nursing women, or women who were of childbearing potential and who were not utilizing an effective contraceptive method. A woman of childbearing potential is defined as a female who is biologically capable of becoming pregnant. Men with partners of childbearing potential not using an effective method of contraception. (Use of effective contraceptives must continue for 3 months after the last dose of everolimus).
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance.
* Uncontrolled diabetes as defined by fasting serum glucose > 2 ULN, severely impaired lung function.
* Cirrhosis/chronic active hepatitis/chronic persistent hepatitis, history of HCV infection (for hepatitis screening indications see section 3.3).
* Drug or alcohol abuse.
* Any other major illness that, in the investigator's judgment, substantially increased the risk associated with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | from 28 days up to 2 years
  Outcome measure in Phase 1 and 2 part
Number of patients progression-free at 4 months. | 4 months
  Outcome measure in phase 2 part
Depletion of circulating CD4+CD25+ regulatory T cells | 28 days
  Treatment schedule that most selectively induces CD4+CD25+ Treg depletion in phase 1 part will be selected for phase 2.

SECONDARY OUTCOMES:
Response rate | 2 years
Frequency of tumor infiltrating CD4+CD25+FOXP3+ regulatory T cells. | 2 years
Peripheral blood drug levels of everolimus and cyclophosphamide | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans J. van der Vliet, MD, PhD, Study Director — Amsterdam UMC, location VUmc
Locations (13):
- Netherlands (13):
  - Medisch Centrum Alkmaar, Alkmaar
  - VU University Medical Center, Amsterdam
  - NKI-AVL, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Ziekenhuis Hoofddorp, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - University Hospital Maastricht, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMC St Radboud Nijmegen, Nijmegen
  - Sint Franciscus Gasthuis Rotterdam, Rotterdam
  - Haga Ziekenhuis, The Hague
  - Medisch Centrum Haaglanden, The Hague
  - Isala Klinieken Zwolle, Zwolle

REFERENCES:
- [Derived] Huijts CM, Werter IM, Lougheed SM, Goedegebuure RS, van Herpen CM, Hamberg P, Tascilar M, Haanen JB, Verheul HM, de Gruijl TD, van der Vliet HJ; Dutch WIN-O Consortium. Phase 1 study of everolimus and low-dose oral cyclophosphamide in patients with metastatic renal cell carcinoma. Cancer Immunol Immunother. 2019 Feb;68(2):319-329. doi: 10.1007/s00262-018-2248-3. Epub 2018 Nov 9. PMID 30413837
- [Derived] Huijts CM, Santegoets SJ, van den Eertwegh AJ, Pijpers LS, Haanen JB, de Gruijl TD, Verheul HM, van der Vliet HJ. Phase I-II study of everolimus and low-dose oral cyclophosphamide in patients with metastatic renal cell cancer. BMC Cancer. 2011 Nov 30;11:505. doi: 10.1186/1471-2407-11-505. PMID 22129044